CLINICAL TRIAL: NCT01171989
Title: Immunogenicity and Safety Study of GlaxoSmithKline Biologicals' GSK2202083A Vaccine Administered as a Booster Dose in 12-18 Months Old Healthy Children
Brief Title: Immunogenicity and Safety Study of GlaxoSmithKline Biologicals' GSK2202083A Vaccine Administered as a Booster Dose
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 113978; 2010-019253-18 (EudraCT Number)
Record Dates: First submitted 2010-07-27; First posted 2010-07-29 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Tetanus; Diphtheria; Haemophilus Influenzae Type b; Hepatitis B; Poliomyelitis; Acellular Pertussis; Diphtheria-Tetanus-aPertussis-Hepatitis B-Poliomyelitis-Haemophilus Influenzae Type b-Neisseria Meni
Keywords: booster vaccination; combined vaccine
MeSH Terms: conditions — Tetanus; Diphtheria; Haemophilus Infections; Hepatitis B; Poliomyelitis | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; PHiD-CV vaccine

ARMS (3):
- GSK2202083A + SYNFLORIX GROUP (Experimental): Healthy male and female subjects between, and including, 12 to 18 months of age at the time of booster vaccination, who were primed with 3 doses of GSK2202083A and Synflorix™ vaccines in the primary study DTPa-HBV-IPV=HIB-MenC-TT-002 (112157), additionally received a booster dose of GSK2202083A vaccine at Day 0 and of Synflorix™ vaccine at Month 1. Both vaccines were administered intramuscularly in the anterolateral side of the thigh.
  Interventions: Biological: GSK2202083A vaccine; Biological: Synflorix™
- INFANRIX HEXA/MENJUGATE GROUP (Active Comparator): Healthy male and female subjects between, and including, 12 to 18 months of age at the time of booster vaccination, who were primed with 3 doses of Infanrix hexa™ vaccine and 2 doses of Menjugate® vaccine in the primary study DTPa-HBV-IPV=HIB-MenC-TT-002 (112157), additionally received a booster dose of Infanrix hexa™ vaccine co-administered with Menjugate® vaccine at Day 0. Both vaccines were administered intramuscularly in the anterolateral side of the thigh.
  Interventions: Biological: Infanrix hexa™; Biological: Menjugate™
- INFANRIX HEXA/NEISVAC-C + SYNFLORIX GROUP (Active Comparator): Healthy male and female subjects between, and including, 12 to 18 months of age at the time of booster vaccination, who were primed with 3 doses of Infanrix hexa™ vaccine and Synflorix™ vaccines in the primary study DTPa-HBV-IPV=HIB-MenC-TT-002 (112157), additionally received a booster dose of Infanrix hexa™ vaccine co-administered with NeisVac-C® vaccine at Day 0 and 1 dose of Synflorix™ vaccine at Month 1. Both vaccines were administered intramuscularly in the anterolateral side of the thigh.
  Interventions: Biological: Infanrix hexa™; Biological: NeisVac-C™; Biological: Synflorix™

INTERVENTIONS:
Biological: GSK2202083A vaccine — Intramuscular, one dose.
  Arms: GSK2202083A + SYNFLORIX GROUP
Biological: Infanrix hexa™ — Intramuscular, one dose.
  Arms: INFANRIX HEXA/MENJUGATE GROUP; INFANRIX HEXA/NEISVAC-C + SYNFLORIX GROUP
Biological: Menjugate™ — Intramuscular, one dose.
  Arms: INFANRIX HEXA/MENJUGATE GROUP
Biological: NeisVac-C™ — Intramuscular, one dose.
  Arms: INFANRIX HEXA/NEISVAC-C + SYNFLORIX GROUP
Biological: Synflorix™ — Intramuscular, one dose.
  Arms: GSK2202083A + SYNFLORIX GROUP; INFANRIX HEXA/NEISVAC-C + SYNFLORIX GROUP

SUMMARY:
The current trial will evaluate the safety and immunogenicity of GSK Biologicals' GSK2202083A vaccine when administered as a booster dose following priming in the first year of life with the same vaccine.

This protocol posting deals with objectives & outcome measures of the booster phase. The objectives & outcome measures of the primary phase are presented in a separate protocol posting (NCT number = NCT00970307).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that parent(s)/ legally acceptable representative(s) can and will comply with the requirements of the protocol.
* Subjects who have completed the full three-dose primary vaccination course according to their group allocation in the primary study DTPa-HBV-IPV=Hib-MenC-TT-002 (112157).
* A male or female between, and including, 12 and 18 months of age at the time of booster vaccination.
* Written informed consent obtained from the parent(s)/ legally acceptable representative(s) of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccines within 30 days preceding the dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the booster vaccination.
* Planned administration/administration of immunoglobulins and/or any blood products within three months before the booster dose, or during the study period.
* Planned administration/administration of any vaccine not foreseen by the study protocol during the period starting 30 days before and ending 30 days after the booster dose.
* Participation in another clinical study since the primary study DTPa-HBV-IPV/Hib-MenC-TT-002 in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Evidence of previous diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis, Hib, pneumococcal and MenC vaccination or disease since the conclusion visit of study DTPa-HBV-IPV/Hib-MenC-TT-002.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* The following adverse event having occurred after previous administration of DTP vaccine:

  * Encephalopathy.
  * Temperature of >= 40.5°C (rectal temperature) within 48 hours of vaccination, not due to another identifiable cause.
  * Collapse or shock-like state within 48 hours of vaccination.
  * Persistent, inconsolable crying occurring within 48 hours of vaccination and lasting >= 3 hours.
  * Seizures with or without fever occurring within 3 days of vaccination.

The following condition is temporary or self-limiting, and a subject may be vaccinated once the condition has resolved if no other exclusion criteria is met:

• Acute disease and/or fever at the time of enrolment.

* Fever is defined as temperature ≥ 37.5°C on oral, axillary or tympanic setting, or ≥ 38.0°C on rectal setting.
* Subjects with a minor illness without fever may be enrolled at the discretion of the investigator.

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 391 (Actual)
Dates: Start 2010-08-18 (Actual); Primary Completion 2010-12-03 (Actual); Study Completion 2010-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- Poland (8):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Dębica
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Siemianowice Śląskie
  - GSK Investigational Site, Tarnów
  - GSK Investigational Site, Torun
  - GSK Investigational Site, Trzebnica
  - GSK Investigational Site, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=137

REFERENCES:
- [Background] Szenborn L, Czajka H, Brzostek J, Konior R, Caubet M, Ulianov L, Leyssen M. A randomized, controlled trial to assess the immunogenicity and safety of a heptavalent diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis, hib and meningococcal serogroup C combination vaccine administered at 2, 3, 4 and 12-18 months of age. Pediatr Infect Dis J. 2013 Jul;32(7):777-85. doi: 10.1097/INF.0b013e31828d6b20. PMID 23838777
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 113978 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113978 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113978 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113978 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113978 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113978 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113978 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Period: Overall Study
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa/Menjugate Group | Infanrix Hexa/NeisVac-C + Synflorix Group
Started | 137 | 133 | 121
Completed | 137 | 133 | 120
Not Completed | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa/Menjugate Group | Infanrix Hexa/NeisVac-C + Synflorix Group | Total
Number analyzed (Participants) | 137 | 133 | 121 | 391
Age, Continuous [Mean (Standard Deviation); unit: Months] | 13.7 (0.71) | 13.8 (0.73) | 13.7 (0.76) | 13.73 (0.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 82 | 56 | 209
  Male | 66 | 51 | 65 | 182
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White-Caucasian/European heritage | 137 | 133 | 121 | 391

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroprotected Subjects Against Polyribosyl-Ribitol-Phosphate (PRP)
Description: A seroprotected subject was defined as a subject with anti-PRP antibody concentrations greater than or equal to (≥) 0.15 micrograms per milliliter (μg/mL).
Time Frame: At Month 1, post-booster dose
Population: The analysis was performed on the Booster According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome variables were available and for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa/Menjugate Group | Infanrix Hexa/NeisVac-C + Synflorix Group
Number analyzed (Participants) | 132 | 126 | 114
Participants | 132 | 126 | 114
Statistical Analysis 1: Comparison: GSK2202083A + Synflorix Group vs Infanrix Hexa/NeisVac-C + Synflorix Group; Difference in percentage anti-PRP ≥ 0.15 μg/mL; Test type: Non-Inferiority — Criterion for evaluation of Non-inferiority: the upper limit of Standardised asymptotic 95% confidence interval lower or equal to 10%; Difference in percentage = 0, 95% CI 2-sided [-3.27 to 2.84]

2. Primary Outcome: Number of Seroprotected Subjects Against Neisseria Meningitidis Serogroup C Using Baby Rabbit Completent (rSBA-MenC)
Description: A seroprotected subject was defined as a subject with anti-rSBA-MenC titers greater than or equal to (≥) 1:8.
Time Frame: At Month 1, post-booster dose
Population: The analysis was performed on the Booster ATP cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome variables were available and for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa/Menjugate Group | Infanrix Hexa/NeisVac-C + Synflorix Group
Number analyzed (Participants) | 131 | 124 | 114
Participants | 131 | 124 | 114
Statistical Analysis 1: Comparison: GSK2202083A + Synflorix Group vs Infanrix Hexa/NeisVac-C + Synflorix Group; Difference between groups for rSBA-MenC ≥1:8; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in percentage = 0, 95% CI 2-sided [-3.27 to 2.86]
Statistical Analysis 2: Comparison: GSK2202083A + Synflorix Group vs Infanrix Hexa/Menjugate Group; Difference between groups for rSBA-MenC ≥1:8; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in percentage = 0, 95% CI 2-sided [-3.02 to 2.86]

3. Secondary Outcome: Number of Seropositive Subjects for Anti-PRP
Description: A seropositive subject was defined as a subject with anti-PRP antibody concentrations ≥ 0.15 μg/mL.
Time Frame: At Month 0, before the booster dose
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa/Menjugate Group | Infanrix Hexa/NeisVac-C + Synflorix Group
Number analyzed (Participants) | 134 | 125 | 113
Participants | 131 | 89 | 88

4. Secondary Outcome: Number of Subjects With Anti-PRP Antibody Concentrations ≥ the Cut-off
Description: The cut-off value of the assay was an anti-PRP antibody concentration ≥ 1 μg/mL.
Time Frame: At Month 0 and Month 1, before and one month after booster dose
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa/Menjugate Group | Infanrix Hexa/NeisVac-C + Synflorix Group
Number analyzed (Participants) | 134 | 126 | 114
Participants
  Anti-PRP, M0: number analyzed (Participants) | 134 | 125 | 113
  Anti-PRP, M0 | 32 | 22 | 15
  Anti-PRP, M1: number analyzed (Participants) | 132 | 126 | 114
  Anti-PRP, M1 | 132 | 126 | 114

5. Secondary Outcome: Anti-PRP Antibody Concentrations
Description: Concentrations were expressed as geometric mean concentrations (GMCs) for the cut-off value of ≥ 0.15 μg/mL.
Time Frame: At Month 0 and Month 1, before and one month after booster dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa/Menjugate Group | Infanrix Hexa/NeisVac-C + Synflorix Group
Number analyzed (Participants) | 134 | 126 | 114
μg/mL
  Anti-PRP, M0: number analyzed (Participants) | 134 | 125 | 113
  Anti-PRP, M0 | 0.601 [0.502 to 0.719] | 0.315 [0.252 to 0.394] | 0.368 [0.302 to 0.449]
  Anti-PRP, M1: number analyzed (Participants) | 132 | 126 | 114
  Anti-PRP, M1 | 25.449 [21.797 to 29.712] | 24.862 [20.188 to 30.619] | 25.943 [21.363 to 31.504]

6. Secondary Outcome: Number of Seroprotected Subjects Against rSBA-MenC
Description: A seroprotected subject was defined as a subject with anti-rSBA-MenC antibody titers ≥ 1:8.
Time Frame: At Month 0, before the booster dose
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa/Menjugate Group | Infanrix Hexa/NeisVac-C + Synflorix Group
Number analyzed (Participants) | 127 | 119 | 104
Participants | 117 | 92 | 10

7. Secondary Outcome: Number of Seropositive Subjects for Anti-rSBA-MenC
Description: A seropositive subject for anti-rSBA-MenC was defined as a subject with antibody titers greater than or equal to (≥) 1:128.
Time Frame: At Month 0 and Month 1, before and one month after booster dose
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa/Menjugate Group | Infanrix Hexa/NeisVac-C + Synflorix Group
Number analyzed (Participants) | 131 | 124 | 114
Participants
  Anti-rSBA-MenC, M0: number analyzed (Participants) | 127 | 119 | 104
  Anti-rSBA-MenC, M0 | 87 | 46 | 3
  Anti-rSBA-MenC, M1 | 130 | 124 | 114

8. Secondary Outcome: Anti-rSBA-MenC Antibody Titres
Description: Antibody titers were expressed as geometric mean titers (GMTs) for the seroprotection cut-off value of ≥ 1:8.
Time Frame: At Month 0 and Month 1, before and one month after booster dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa/Menjugate Group | Infanrix Hexa/NeisVac-C + Synflorix Group
Number analyzed (Participants) | 131 | 124 | 114
Titers
  Anti-rSBA-MenC, M0: number analyzed (Participants) | 127 | 119 | 104
  Anti-rSBA-MenC, M0 | 148.8 [114.4 to 193.5] | 55.6 [40.8 to 75.6] | 5.4 [4.5 to 6.6]
  Anti-rSBA-MenC, M1 | 2703.4 [2289.6 to 3192.1] | 7701.8 [6511.9 to 9109] | 2320.4 [2040.3 to 2638.8]

9. Secondary Outcome: Number of Subjects With Polysaccharide N. Meningitidis Serogroup C (PSC) Antibody Concentrations ≥ Cut-off Values
Description: The cut-off values assessed were ≥ 0.3 μg/mL and ≥ 2 μg/mL.
Time Frame: At Month 0 and Month 1, before and one month after booster dose
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa/Menjugate Group | Infanrix Hexa/NeisVac-C + Synflorix Group
Number analyzed (Participants) | 134 | 126 | 114
Participants
  Anti-PSC ≥ 0.3 μg/mL, M0 | 133 | 101 | 0
  Anti-PSC ≥ 0.3 μg/mL, M1: number analyzed (Participants) | 134 | 125 | 114
  Anti-PSC ≥ 0.3 μg/mL, M1 | 134 | 125 | 114
  Anti-PSC ≥ 2 μg/mL, M0 | 72 | 21 | 0
  Anti-PSC ≥ 2 μg/mL, M1: number analyzed (Participants) | 134 | 125 | 114
  Anti-PSC ≥ 2 μg/mL, M1 | 129 | 125 | 114

10. Secondary Outcome: Anti-PSC Antibody Concentrations
Description: Concentrations were expressed as geometric mean concentrations (GMCs) for the seropositivity cut-off value of ≥ 0.3 μg/mL.
Time Frame: At Month 0 and Month 1, before and one month after booster dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa/Menjugate Group | Infanrix Hexa/NeisVac-C + Synflorix Group
Number analyzed (Participants) | 134 | 126 | 114
μg/mL
  Anti-PSC, M0 | 1.98 [1.69 to 2.31] | 0.76 [0.63 to 0.91] | 0.15 [0.15 to 0.15]
  Anti-PSC, M1: number analyzed (Participants) | 134 | 125 | 114
  Anti-PSC, M1 | 6.91 [6.21 to 7.69] | 21.75 [18.9 to 25.04] | 17.7 [15.97 to 19.61]

11. Secondary Outcome: Number of Seropositive Subjects for Anti-diphteria (Anti-D) and Anti-tetanus (Anti-T)
Description: A seropositive subject was defined as a subject with anti-D and anti-T antibody concentrations ≥ 0.1 international units per milliliter (IU/mL).
Time Frame: At Month 0 and Month 1, before and one month after booster dose
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa/Menjugate Group | Infanrix Hexa/NeisVac-C + Synflorix Group
Number analyzed (Participants) | 134 | 126 | 114
Participants
  Anti-D, M0: number analyzed (Participants) | 134 | 125 | 113
  Anti-D, M0 | 129 | 115 | 108
  Anti-D, M1: number analyzed (Participants) | 132 | 126 | 114
  Anti-D, M1 | 132 | 126 | 114
  Anti-T, M0: number analyzed (Participants) | 134 | 125 | 112
  Anti-T, M0 | 133 | 118 | 111
  Anti-T, M1: number analyzed (Participants) | 132 | 126 | 114
  Anti-T, M1 | 132 | 126 | 114

12. Secondary Outcome: Anti-D and Anti-T Antibody Concentrations
Description: Concentrations were expressed as geometric mean concentrations (GMCs) for the seropositivity cut-off value of ≥ 0.1 IU/mL.
Time Frame: At Month 0 and Month 1, before and one month after booster dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa/Menjugate Group | Infanrix Hexa/NeisVac-C + Synflorix Group
Number analyzed (Participants) | 134 | 126 | 114
IU/mL
  Anti-D, M0: number analyzed (Participants) | 134 | 125 | 113
  Anti-D, M0 | 0.349 [0.308 to 0.395] | 0.316 [0.27 to 0.37] | 0.311 [0.274 to 0.354]
  Anti-D, M1: number analyzed (Participants) | 132 | 126 | 114
  Anti-D, M1 | 6.166 [5.47 to 6.951] | 7.351 [6.63 to 8.15] | 6.02 [5.367 to 6.752]
  Anti-T, M0: number analyzed (Participants) | 134 | 125 | 112
  Anti-T, M0 | 0.895 [0.808 to 0.992] | 0.316 [0.275 to 0.365] | 0.567 [0.5 to 0.643]
  Anti-T, M1: number analyzed (Participants) | 132 | 126 | 114
  Anti-T, M1 | 11.945 [10.898 to 13.094] | 5.351 [4.752 to 6.027] | 11.638 [10.398 to 13.025]

13. Secondary Outcome: Number of Subjects With Anti-hepatitis B (Anti-HBs) Antibody Concentrations ≥ Cut-off Values
Description: The cut-off values assessed were 3.3 milli-international units per milliliter (mIU/mL), 10 mIU/mL and 100 mIU/mL.
Time Frame: At Month 0 and Month 1, before and one month after booster dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa/Menjugate Group | Infanrix Hexa/NeisVac-C + Synflorix Group
Number analyzed (Participants) | 125 | 122 | 111
Participants
  Anti-HBs ≥ 3.3 mIU/mL, M0: number analyzed (Participants) | 124 | 122 | 105
  Anti-HBs ≥ 3.3 mIU/mL, M0 | 123 | 120 | 104
  Anti-HBs ≥ 10 mIU/mL, M0: number analyzed (Participants) | 124 | 122 | 105
  Anti-HBs ≥ 10 mIU/mL, M0 | 121 | 119 | 102
  Anti-HBs ≥ 100 mIU/mL, M0: number analyzed (Participants) | 124 | 122 | 105
  Anti-HBs ≥ 100 mIU/mL, M0 | 99 | 108 | 90
  Anti-HBs ≥ 3.3 mIU/mL, M1: number analyzed (Participants) | 125 | 114 | 111
  Anti-HBs ≥ 3.3 mIU/mL, M1 | 125 | 114 | 111
  Anti-HBs ≥ 10 mIU/mL, M1: number analyzed (Participants) | 125 | 114 | 111
  Anti-HBs ≥ 10 mIU/mL, M1 | 125 | 114 | 109
  Anti-HBs ≥ 100 mIU/mL, M1: number analyzed (Participants) | 125 | 114 | 111
  Anti-HBs ≥ 100 mIU/mL, M1 | 123 | 113 | 109

14. Secondary Outcome: Anti-HBs Antibody Concentrations
Description: Concentrations were presented as geometric mean concentrations (GMCs), expressed in mIU/mL.
Time Frame: At Month 0 and Month 1, before and after booster dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa/Menjugate Group | Infanrix Hexa/NeisVac-C + Synflorix Group
Number analyzed (Participants) | 125 | 122 | 111
mIU/mL
  Anti-HBs, M0: number analyzed (Participants) | 124 | 122 | 105
  Anti-HBs, M0 | 295.1 [234 to 372.1] | 387.6 [302.6 to 496.3] | 330.4 [256.5 to 425.5]
  Anti-HBs, M1: number analyzed (Participants) | 125 | 114 | 111
  Anti-HBs, M1 | 6390.7 [5171.5 to 7897.2] | 8465 [6827 to 10496.1] | 6840.3 [5235.8 to 8936.6]

15. Secondary Outcome: Number of Seropositive Subjects for Anti-poliovirus Types 1, 2 and 3
Description: A seropositive subject was defined as a subject with anti-polio type 1, 2 or 3 ≥ 1:8.
Time Frame: At Month 0 and Month 1, before and one month after booster dose
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa/Menjugate Group | Infanrix Hexa/NeisVac-C + Synflorix Group
Number analyzed (Participants) | 113 | 102 | 95
Participants
  Anti-polio 1, M0: number analyzed (Participants) | 103 | 101 | 88
  Anti-polio 1, M0 | 96 | 96 | 79
  Anti-polio 1, M1: number analyzed (Participants) | 113 | 99 | 94
  Anti-polio 1, M1 | 113 | 99 | 94
  Anti-polio 2, M0: number analyzed (Participants) | 104 | 100 | 88
  Anti-polio 2, M0 | 93 | 95 | 80
  Anti-polio 2, M1: number analyzed (Participants) | 113 | 100 | 94
  Anti-polio 2, M1 | 113 | 100 | 94
  Anti-polio 3, M0: number analyzed (Participants) | 102 | 102 | 88
  Anti-polio 3, M0 | 94 | 94 | 80
  Anti-polio 3, M1: number analyzed (Participants) | 113 | 100 | 95
  Anti-polio 3, M1 | 113 | 100 | 95

16. Secondary Outcome: Anti-poliovirus Types 1, 2 and 3 Antibody Titres
Description: Titers were expressed as geometric mean titters (GMTs) for the seropositivity cut-off value of ≥ 1:8.
Time Frame: At Month 0 and Month 1, before and one month after booster dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa/Menjugate Group | Infanrix Hexa/NeisVac-C + Synflorix Group
Number analyzed (Participants) | 113 | 102 | 95
Titers
  Anti-polio 1, M0: number analyzed (Participants) | 103 | 101 | 88
  Anti-polio 1, M0 | 35.1 [27.8 to 44.4] | 48.3 [37.3 to 62.6] | 37 [28.5 to 48]
  Anti-polio 1, M1: number analyzed (Participants) | 113 | 99 | 94
  Anti-polio 1, M1 | 870.5 [721.5 to 1050.2] | 1203 [982.3 to 1473.2] | 896.7 [739.1 to 1088]
  Anti-polio 2, M0: number analyzed (Participants) | 104 | 100 | 88
  Anti-polio 2, M0 | 34.9 [27.6 to 44.2] | 46.2 [35.2 to 60.8] | 38.2 [29.2 to 50.1]
  Anti-polio 2, M1: number analyzed (Participants) | 113 | 100 | 94
  Anti-polio 2, M1 | 1179.1 [979.3 to 1419.7] | 1483.6 [1217.2 to 1808.5] | 1143.8 [929.7 to 1407.1]
  Anti-polio 3, M0: number analyzed (Participants) | 102 | 102 | 88
  Anti-polio 3, M0 | 43.7 [34 to 56.1] | 51.6 [39.6 to 67.1] | 48.5 [36.3 to 64.7]
  Anti-polio 3, M1: number analyzed (Participants) | 113 | 100 | 95
  Anti-polio 3, M1 | 1493.3 [1195 to 1866] | 1832.9 [1507.9 to 2228.1] | 1416.8 [1157.1 to 1734.8]

17. Secondary Outcome: Number of Seropositive Subjects for Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN)
Description: A seropositive subject was defined as a subject with anti-PT, anti-FHA and anti-PRN antibody concentrations ≥ 5 enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: At Month 0 and Month 1, before and one month after booster dose
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa/Menjugate Group | Infanrix Hexa/NeisVac-C + Synflorix Group
Number analyzed (Participants) | 133 | 126 | 114
Participants
  Anti-PT, M0: number analyzed (Participants) | 133 | 125 | 112
  Anti-PT, M0 | 98 | 97 | 84
  Anti-PT, M1 | 133 | 126 | 114
  Anti-FHA, M0: number analyzed (Participants) | 132 | 125 | 112
  Anti-FHA, M0 | 131 | 122 | 111
  Anti-FHA, M1: number analyzed (Participants) | 132 | 126 | 114
  Anti-FHA, M1 | 132 | 126 | 114
  Anti-PRN, M0: number analyzed (Participants) | 133 | 126 | 113
  Anti-PRN, M0 | 100 | 109 | 94
  Anti-PRN, M1: number analyzed (Participants) | 132 | 126 | 113
  Anti-PRN, M1 | 132 | 126 | 113

18. Secondary Outcome: Anti-PT, Anti-FHA and Anti-PRN Antibody Concentrations
Description: Concentrations were expressed as geometric mean concentrations (GMCs) for the seropositivity cut-off value ≥ 5 EL.U/mL.
Time Frame: At Month 0 and Month 1, before and one month after booster dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa/Menjugate Group | Infanrix Hexa/NeisVac-C + Synflorix Group
Number analyzed (Participants) | 133 | 126 | 114
EL.U/mL
  Anti-PT, M0: number analyzed (Participants) | 133 | 125 | 112
  Anti-PT, M0 | 7.7 [6.7 to 8.8] | 8.9 [7.7 to 10.2] | 7.1 [6.2 to 8.1]
  Anti-PT, M1 | 50.6 [45.1 to 56.7] | 66.3 [58.6 to 75] | 61.8 [53.7 to 71.1]
  Anti-FHA, M0: number analyzed (Participants) | 132 | 125 | 112
  Anti-FHA, M0 | 24.3 [21 to 28.2] | 30.4 [26.2 to 35.4] | 25.7 [22.1 to 29.7]
  Anti-FHA, M1: number analyzed (Participants) | 132 | 126 | 114
  Anti-FHA, M1 | 265.3 [235.3 to 299] | 339.6 [300.2 to 384.1] | 325.2 [284.7 to 371.4]
  Anti-PRN, M0: number analyzed (Participants) | 133 | 126 | 113
  Anti-PRN, M0 | 8.8 [7.5 to 10.3] | 12.7 [10.9 to 14.9] | 11 [9.3 to 13]
  Anti-PRN, M1: number analyzed (Participants) | 132 | 126 | 113
  Anti-PRN, M1 | 216.8 [183.7 to 255.8] | 319.8 [275.6 to 371.2] | 277.9 [233.1 to 331.4]

19. Secondary Outcome: Number of Subjects With Any Solicited Local Symptoms
Description: Solicited local symptoms assessed included pain, redness and swelling. Any= all reports of the speecified symptom irrespective of intensity grade.
Time Frame: During the 8-day (Days 0-7) post-booster period
Population: The analysis was performed on the Booster Total Vaccinated Cohort, which included all subjects with the booster vaccine administration documented and who had the symptoms sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa/Menjugate Group | Infanrix Hexa/NeisVac-C + Synflorix Group
Number analyzed (Participants) | 136 | 133 | 120
Participants
  Any Pain | 44 | 68 | 58
  Any Redness | 69 | 77 | 69
  Any Swelling | 50 | 58 | 50

20. Secondary Outcome: Number of Subjects With Any Solicited General Symptoms
Description: Solicited general symptoms assessed included drowsiness, irritability, loss of appetite and fever (defined as axillary temperature ≥ 37.5º C). Any= all reports of the specified symptom irrespective of intensity grade and relationship to vaccination.
Time Frame: During the 8-day (Days 0-7) post-booster period
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa/Menjugate Group | Infanrix Hexa/NeisVac-C + Synflorix Group
Number analyzed (Participants) | 136 | 133 | 120
Participants
  Any Drowsiness | 40 | 39 | 39
  Any Irritability | 65 | 65 | 66
  Any Loss of appetite | 31 | 32 | 43
  Any Temperature (Axillary) | 34 | 30 | 31

21. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE was any AE (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: During the 31-day (Days 0-30) post-booster period
Population: The analysis was performed on the Booster Total Vaccinated Cohort, which included all subjects with the booster vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa/Menjugate Group | Infanrix Hexa/NeisVac-C + Synflorix Group
Number analyzed (Participants) | 137 | 133 | 121
Participants | 45 | 29 | 35

22. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs were defined as medical occurrences that resulted in death, were life threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity.
Time Frame: After the booster dose of the study vaccine up to the study end (from Month 0 to Month 1)
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa/Menjugate Group | Infanrix Hexa/NeisVac-C + Synflorix Group
Number analyzed (Participants) | 137 | 133 | 121
Participants | 3 | 2 | 2

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 8-day (Days 0- 7) post-booster vaccination. Unsolicited adverse events: during the 31-day (Days 0- 30) post-booster vaccination. Serious adverse events: entire booster period (from Month 0 up to Month 1).
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa/Menjugate Group | Infanrix Hexa/NeisVac-C + Synflorix Group
All-Cause Mortality (participants affected / at risk) | 0/137 | 0/133 | 0/121
Serious Adverse Events (participants affected / at risk) | 3/137 | 2/133 | 2/121
Other Adverse Events (participants affected / at risk) | 114/137 | 114/133 | 102/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2202083A + Synflorix Group (N=137) | Infanrix Hexa/Menjugate Group (N=133) | Infanrix Hexa/NeisVac-C + Synflorix Group (N=121)
Thermal burn (Injury, poisoning and procedural complications) | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | GSK2202083A + Synflorix Group (N=137) | Infanrix Hexa/Menjugate Group (N=133) | Infanrix Hexa/NeisVac-C + Synflorix Group (N=121)
Pain (General disorders) | 44/136 | 68 | 58/120 — This solicited local symptom was only collected from subjects with their symptom sheets completed.
Redness (General disorders) | 69/136 | 77 | 69/120 — This solicited local symptom was only collected from subjects with their symptom sheets completed.
Swelling (General disorders) | 50/136 | 58 | 50/120 — This solicited local symptom was only collected from subjects with their symptom sheets completed.
Drowsiness (General disorders) | 40/136 | 39 | 39/120 — This solicited general symptom was only collected from subjects with their symptom sheets completed.
Irritability (General disorders) | 65/136 | 65 | 66/120 — This solicited general symptom was only collected from subjects with their symptom sheets completed.
Loss of appetite (General disorders) | 31/136 | 32 | 43/120 — This solicited general symptom was only collected from subjects with their symptom sheets completed.
Fever (General disorders) | 34/136 | 30 | 31/120 — This solicited general symptom was only collected from subjects with their symptom sheets completed.
Upper respiratory tract infection (unsolicited) (Infections and infestations) | 6 | 11 | 6
Rhinitis (Infections and infestations) | 9 | 4 | 8
Nasopharyngitis (Infections and infestations) | 7 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.